CLINICAL TRIAL: NCT04048408
Title: Assessment of Cognitive Status, Pain, Functional Status, Postural Awareness, Respiratory Muscle Strength and Endurance in Obstructive Pulmonary Diseases
Brief Title: Comparison of Respiratory Muscle, Pain, Functional Performance and Cognitive Status in Obstructive Lung Diseases
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Naciye Vardar-Yagli, Associate Professor, Hacettepe University
Other Study IDs: GO 18/109
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Pain, Chronic; Obstructive Pulmonary Disease; Cognitive Impairment; Functional Disturbance
MeSH Terms: conditions — Chronic Pain; Lung Diseases, Obstructive; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obstructive lung diseases group
- Healthy group

SUMMARY:
In the literature, there are a limited number of studies evaluating postural awareness, cognitive status, respiratory muscle strength and endurance, functional capacity, and pain in people with obstructive pulmonary disease, and comparing these parameters with each other and with healthy subjects, and most of the studies are on chronic obstructive pulmonary disease patients. There we will evaluate these parameters in different obstructive lung diseases and compare the findings of healthy individuals.

ELIGIBILITY:
Inclusion Criteria for obstructive lung diseases

1. To be diagnosed with obstructive pulmonary disease,
2. Have not experienced acute exacerbation in the last 3 months,
3. Being between the ages of 18-65,
4. Not having chronic pain problems,
5. Volunteer for research,
6. To be able to walk and cooperate.

Exclusion criteria for obstructive lung diseases

1. To be able to diagnose neurological disorder,
2. To have an advanced orthopedic disease that may affect functional capacity measurement.

Criteria for Non-Inclusion for healthy group

1. To have any cardiopulmonary disease,
2. To have an advanced orthopedic disease that may affect functional capacity measurement.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obstructive lung diseases in 18-65 years old
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
Pain Perception | 01.01.2019-31.08.2019
  Pain Perception Threshold and Tolerance With Algometer

SECONDARY OUTCOMES:
Cognitive Function Assessment | 01.01.2019-31.08.2019
  Montreal Cognitive Assessment Test (MoCA)
Functional capacity assesment | 01.01.2019-31.08.2019
  6 minute walk test
Postural awareness assesment | 01.01.2019-31.08.2019
  Body Awareness Questionnare is a likert type questionnare and total score ranges from 18-126. Higher scores mean better body awareness level
Respiratory muscle strength and endurance measurement | 01.01.2019-31.08.2019
  Mouth pressure measurement

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Calik Kutukcu, PhD, Principal Investigator — Hacettepe University; Melda Saglam, PhD, Principal Investigator — Hacettepe University; Deniz Inal Ince, Professor, Principal Investigator — Hacettepe University; Hulya Arikan, Professor, Principal Investigator — Hacettepe University; Naciye Vardar Yagli, PhD, Study Director — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Ankara, Please Choose A State, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No